CLINICAL TRIAL: NCT01201746
Title: Influence of Periodontal Treatment on Systemic Inflammatory Mediators:hsC-reactive Protein, Fibrinogen and White Blood Cells in CHD Patients
Brief Title: Influence of Periodontal Treatment on Systemic Inflammatory Mediators
Acronym: Perio-CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Collaborators: Higher Education Commission (Pakistan) (Other)
Responsible Party: Principal Investigator, Syed Akhtar Hussain Bokhari, PhD Candidate, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PU-D/314/Acad; HEC-20-685/06 (Other Grant/Funding Number: Higher Education Commission, Govt of Pakistan, Islamabad)
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2010-09

CONDITIONS: Periodontal Disease; Coronary Heart Disease
Keywords: Non-surgical periodontal therapy; Coronary heart disease (CHD); periodontal Disease; hsCRP; Fibrinogen; WBCs
MeSH Terms: conditions — Periodontal Diseases; Coronary Disease | interventions — Treatment Delay; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Periodontal Therapy (Experimental): Scaling Root planing and oral hygiene instructions
  Interventions: Procedure: Periodontal therapy
- Delayed treatment (Placebo Comparator): Scaling Root planing and oral hygiene instructions
  Interventions: Procedure: Delayed treatment

INTERVENTIONS:
Procedure: Delayed treatment — Scaling, Root Planing and oral hygiene instruction
  Other Names: Control group
  Arms: Delayed treatment
Procedure: Periodontal therapy — Scaling, root planning and oral hygiene instructions
  Other Names: Experimental group
  Arms: Periodontal Therapy

SUMMARY:
Currently the research issue in establishing the role of periodontal disease (PD) in coronary heart disease (CHD) risk is to define the pathways that lead to cause-effect relationship between PD and CHD. There is no consensus on definition of a periodontal disease case or the threshold level that may give clear indication for this relationship. Periodontal therapy has been used in different studies with the hope that a change in periodontal disease status may modify the factors associated with CHD risk. Many of these studies, on role of periodontal therapy in the reduction of CHD associated risk-factors, were based on small study samples, and very few studies were randomized controlled trials. So a need for large prospective studies is warranted in literature.----------- A single-blind parallel-arm randomized controlled clinical trial was designed to observe the influence of periodontal treatment on serum inflammatory mediators of hsC-reactive protein, white blood cells and fibrinogen in CHD patients.

Hypothesis: Periodontal therapy in CHD patients, by reducing periodontal inflammation, may decrease the host systemic inflammatory burden associated with atherogenic processes.

ELIGIBILITY:
Inclusion Criteria:

A. General/Medical

1. Any race/ethnic group
2. Aged > 30 years
3. Male or female
4. CHD case (CHD angiographically confirmed)
5. CHD diagnosed > 3 months prior to entry into study.
6. No acute or chronic systemic conditions (see exclusion criteria below)
7. No medications/medication history that can interfere with the study (see exclusion criteria below)
8. Non-smoker (=Never smoker) or former smoker (=Does not smoke now and has not smoked at all for a minimum of the last 12 consecutive months)
9. Able and willing to comply with study procedures
10. Able and willing to be available for the duration of the study
11. Able and willing to provide signed informed consent

B. Oral/Periodontal

1. Dentate with at least 14 natural teeth, excluding third molars, that can be evaluated periodontally.
2. Baseline whole mouth BOP > 20% of sites.
3. Periodontitis case; periodontitis case defined as subject having ≥ 4 teeth with ≥ 1 site with PPD ≥ 4 mm & CAL ≥ 3 mm at same site
4. No mechanical periodontal therapy in the last 6 months.
5. No acute oral diseases (mucosal lesions), oral infections, need for immediate dental/periodontal care (e.g., NUG).

Exclusion Criteria:

A. General/Medical

1. Age ≤ 30 years
2. Not fulfilling criteria of defined CHD case
3. Fulfilling criteria of defined CHD case, but diagnosed ≤ 3 months prior to start of study
4. Current smoker
5. Former smoker who does not smoke but who has smoked ≥ 1 cigarette (or equivalent, in form of water pipe, pipe, cigar) in the last 12 months.
6. Females pregnant or lactating
7. Systemic chronic conditions known to be associated with periodontitis or with changes in systemic inflammation: Diabetes,Rheumatoid Arthritis, Rheumatic Fever, SLE, Malignancy, Respiratory diseases, Renal diseases, Other (e.g., autoimmune diseases, fungal infections, immunological deficiencies, etc.)
8. Systemic acute conditions known to affect systemic markers of inflammation: Acute bacterial infection, Acute viral infection (common cold, influenza, sinusitis), Orthopedic trauma, Surgery
9. Medications known to affect systemic inflammatory biomarkers: Statins, Systemic steroids, Non-steroidal anti-inflammatory drugs, Immunosuppressants,
10. Medications potentially affecting systemic inflammatory markers, if therapy started less than 3 months prior to study such as Hormone replacement therapy, Contraceptives
11. Systemic antibiotic therapy in the last 3 months
12. Unable or unwilling to comply with study procedures
13. Unable or unwilling to be available for the duration of the study
14. Unable or unwilling to provide signed informed consent

B. Oral/Periodontal

1. <14 teeth that can be periodontally evaluated (excluding 3rd molars)
2. BOP ≤ 20% of sites
3. Not fulfilling criteria of defined periodontitis case
4. Having received any periodontal therapy within last 6 months
5. Topical/local antibiotic or anti-inflammatory therapy in last 6 months
6. Acute oral infections
7. Oral wounds, including recent (< 2 months) extractions

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
high-sensitivity C-Reactive Protein (hsCRP) | 1-3 months

SECONDARY OUTCOMES:
Fibrinogen | 1-3 months
White Blood Cells | 1-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ayyaz A Khan, Ph.D., Study Director — Sheikh Zayed Federal Postgraduate Medical Institute; Syed Akhtar H Bokhari, MCPS, Principal Investigator — Sheikh Zayed Federal Postgraduate Medical Institute; Mohammad Azhar, MRCP, Study Chair — Punjab Institute of Cardiology
Locations (1):
- Punjab Institute of Cardiology, Lahore, Punjab Province, Pakistan